CLINICAL TRIAL: NCT01271842
Title: Long-term Outcome and Lung Capacity in Survivors of ARDS Due to Influenza A (H1N1) v2009 The RESPIFLU Study
Acronym: RESPIFLU
Status: Completed | Type: Observational
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: C10-26; 2010-A00741-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2025-10-07 (Actual); Status verified 2012-12

CONDITIONS: Influenza; Pneumonia, Viral; Pulmonary Fibrosis; Quality of Life; Stress Disorders, Post Traumatic
MeSH Terms: conditions — Influenza, Human; Pneumonia, Viral; Pulmonary Fibrosis; Combat Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Extra corporeal oxygenation: Survivors of ARDS due to influenza A (H1N1)2009 infection who needed an extracorporeal oxygenation at the time of infection
- No extracorporeal oxygenation: Survivors of ARDS due to influenza A (H1N1) 2009 infection who did not need an extracorporeal oxygenation at the time of infection

SUMMARY:
Influenza A (H1N1) v2009 infection was responsible throughout the world of viral pneumonia and severe pulmonary edema requiring rescue therapeutics such as extracorporeal oxygenation. To date, no data exist on the outcome of patients having developed acute respiratory distress syndrome (ARDS) due to influenza A (H1N1) v2009, and in particular in patients with very severe lung injury requiring extracorporeal oxygenation. Although data exist on long-term outcome of survivors of ARDS, the patients included in the observational studies were heterogeneous with various underlying disease. Moreover, no study compared the outcome of survivors of ARDS according to the need or not of extracorporeal oxygenation. We therefore conducted this prospective case-control study to compare the long term pulmonary and extra pulmonary function in 2 groups of patients, one with severe ARDS due to H1N1 requiring extracorporeal oxygenation (case), and the second with ARDS due to H1N1 but without need for extracorporeal oxygenation (control). Eighteen case patients with inclusion and without non-inclusion criteria were selected from our national registry, and 32 controls (with inclusion and exclusion criteria) were matched on age, sex, and body mass index. All 48 patients will be contacted and asked to participate. Patients will be evaluate at least 9 months after ICU discharge, looking for health-related quality of life, measured by the Medical Outcomes Study 36-item Short-Form General Health Survey (SF-36), post traumatic stress disorder, assessed by the Impact of Event Scale Anxiety, and depression, assessed by the Hospital and Depression Score. Pulmonary function testing, including VO2 max test on a static bike will be performed. Muscle weakness will be clinically evaluated by the medical council research (MRC) test, with an additional electromyography if the result of the test was <48/60. A CT-scan will be performed, looking for lung abnormalities (fibrosis...). Albumin and prealbumin will be measured to evaluate the nutritional status.

Primary outcome measurement is carbon monoxide diffusion capacity. The primary hypothesis is that patients with extracorporeal oxygenation will have a carbon monoxide diffusion capacity lower than patients without extracorporeal oxygenation (15% difference between groups). Inclusion of 13 patients in the case group and 26 patients in the control group will allow testing this hypothesis with a statistical power of 80% (standard deviation 15%). Secondary outcome measures will be the quality of life, the presence or not of post-traumatic stress disorders, of anxiety and/or depression, the results of pulmonary function testing, of the CT-scan, and of muscle testing. All results will be compared in patients with and without extracorporeal oxygenation.

ELIGIBILITY:
Inclusion Criteria:

* Patients from 18 to 65 year-old
* Survivors of ARDS due to influenza A (H1N1) v2009 infection developed during the winter 2009-2010
* Influenza A (H1N1) infection confirmed by RT-PCR
* Written consent
* Need or not for extra corporeal lung oxygenation

Exclusion Criteria:

* Pre existing pulmonary disease
* Asthma
* Diabetes mellitus
* Immunodepression
* Cancer
* Severe obesity (BMI >35 kg/m²)
* Neuromuscular disease
* Pre existing cardiac disease
* Chronic renal failure
* Liver failure
* Stroke
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two groups of survivors of severe acute respiratory distress syndrome due to influenza A H1N1 infection will be recruited; the first required extracorporeal oxygenation at the time of viral infection, and the second did not require extracorporeal oxygenation at the time of viral infection. Patients will be recruited at least 9 months after ICU discharge. Eighteen case patients matching inclusion and non-inclusion criteria were selected from our national registry, and 32 controls (with inclusion and exclusion criteria) were matched on age, sex, and body mass index.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2011-10-02 (Actual); Study Completion 2011-10-02 (Actual)

PRIMARY OUTCOMES:
Carbon monoxide diffusion capacity | At least 9 months after ICU discharge

SECONDARY OUTCOMES:
Health-related quality of life | At least 9 months after ICU discharge
Pulmonary function testing | At least 9 months after ICU discharge
Post traumatic stress disorder | At least 9 months after ICU discharge
Anxiety and depression | At least 9 months after ICU discharge
Muscle weakness | At least 9 months after ICU discharge
Lung abnormalities on CT scan | At least 9 months after ICU discharge
Alveoli-arterial gradient of oxygen during effort | At least 9 months after ICU discharge

CONTACTS AND LOCATIONS:
Overall Officials: Charles-Edouard Luyt, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- CHU Pitié-Salpêtrière, Paris, France

REFERENCES:
- [Result] Luyt CE, Combes A, Becquemin MH, Beigelman-Aubry C, Hatem S, Brun AL, Zraik N, Carrat F, Grenier PA, Richard JM, Mercat A, Brochard L, Brun-Buisson C, Chastre J; REVA Study Group. Long-term outcomes of pandemic 2009 influenza A(H1N1)-associated severe ARDS. Chest. 2012 Sep;142(3):583-592. doi: 10.1378/chest.11-2196. PMID 22948576